CLINICAL TRIAL: NCT03020732
Title: Concentrated Growth Factor Membrane Versus Subepithelial Connective Tissue Grafts in Treatment of Multiple Gingival Recession Defects: a Split-mouth Randomized Clinical Trial
Brief Title: Gingival Recession Treatment With Concentrated Growth Factor(CGF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, serap karakış akcan, phd doctor, Gazi University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03/2011-16
Record Dates: First submitted 2016-12-30; First posted 2017-01-13 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Gingival Recession
Keywords: growth factor; mucogingival surgery; gingival recession
MeSH Terms: conditions — Gingival Recession | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- test groups (Experimental): In this split mouth study, bilaterally gingival recession defects were randomly treated in test(CGF+CAF) or control(SCTG+CAF) groups.In test groups, a special centrifuge machine(Medifuge) and subjects venous blood were used to obtain Concentrated growth factor. A special compress was used to transform Concentrated growth factor membrane.
  Interventions: Procedure: test groups
- control groups (Active Comparator): In this split mouth study, bilaterally gingival recession defects were randomly treated in test(CGF+CAF) or control(SCTG+CAF) groups. In control groups, subepithelial connective tissue graft was taken from the palatal canine teeth-first molar teeth area with a trap door technique according to the width of the exposed root surface and the adjacent bone margins. The graft's thickness was adjusted between 1.5 and 2 mm.
  Interventions: Procedure: control groups

INTERVENTIONS:
Procedure: test groups — Coronally advanced flap procedure is a mucogingival surgery technique that was used to prepare recipient sites. Concentrated growth factor(CGF) membranes were placed over the exposed root surface. The flap was advanced 1 mm coronally from CEJ to completely cover.
  Other Names: CGF+ CAF groups
  Arms: test groups
Procedure: control groups — Coronally advanced flap procedure is a mucogingival surgery technique that was used to prepare recipient sites. Subepithelial connective tissue graft was placed over the exposed root surface. The flap was advanced 1 mm coronally from CEJ to completely cover.
  Other Names: SCTG+CAF
  Arms: control groups

SUMMARY:
Platelet concentrates(PC) are used in the field of periodontology and implantology for the content necessary key cells and growth factors to accelerate healing and to provide regeneration. Concentrated Growth Factors(CGF) is defined as an innovative method or a new generation PC. The purpose of this clinical study was to evaluate the clinical effectiveness of Concentrated Growth Factor(CGF) membrane with coronally advanced flap(CAF) procedure's and subepithelial connective tissue graft(SCTG) with CAF in the treatment of Miller class I gingival recessions (GR).

DETAILED DESCRIPTION:
CGF is defined as an innovative method to produce platelet rich fibrin(PRF) or a new generation platelet concentrate(PC).The rotational speed of the centrifuge machine used in CGF, varies between 2400-3000 rpm. The variability of the rotation speed during centrifugation allows a fibrin matrix that larger, more intensive and includes more growth factors than PRF. Some studies have been reported that CGF have an inducing effect on periodontal ligament stem cells for osteogenic differentiation and clinically provides new bone formation for the sinus augmentation. In literature, there is only one clinical research associated with multiple gingival recession defects treatment. It showed that CGF with CAF surgery increases keratinized gingiva weight and thickness and it maybe prevents post-operative relapse for CAF.

PC has also been mentioned to be effective in to increase the width of keratinized tissue with providing root coverage and it may reduce early post-surgical complications, and accelerate wound healing in systematic review. In the treatment of isolated or multiple gingival recession, PRF and SCTG with CAF procedures have been reported to similar root coverage. PRF can be used as an alternative method for SCTG .CGF and PRF have similar composition. However higher resistance and viscosity of CGF may protect growth factors from proteolysis better than PRF. There is any comparative study for CGF and SCTG in literature in terms of clinically or patient related parameters.

Therefore, the purpose of this clinical study is to evaluate the clinical efficacy of CGF in combination with CAF in the treatment of gingival recession's defects, and to compare SCTG in combination with CAF. It is also aimed to asses and compare postoperative pain and soft tissue healing.

ELIGIBILITY:
Inclusion Criteria:

* age≥18
* systemically and periodontally healthy non-smoker patients
* multiple, adjacent, bilaterally Miller class I
* recession depth ≥2 and ≤5 mm, probing depth≤3 mm, located lateral, canine or premolars on same arch(maxilla or mandibula)
* identifiable cemento-enamel junction
* absence caries or restoration on buccal surface, endodontic treatment or problem
* palatal donor tissue thickness ≥3 mm for SCTG

Exclusion Criteria:

* patients have smoking habit or systemic diseases that might be contraindication for periodontal surgery
* the presence of using medication affect that blood clotting mechanism and wound healing
* previous periodontal surgeries in gingival recession areas
* pregnancy, lactation,or oral contraceptive drug intake for female patients
* insufficient oral hygiene (full- mouth plaque and bleeding scores ≥15% after phase I periodontal treatment)
* unchanged traumatic tooth-brushing habit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
recession depth | change from baseline at following surgery first, third and sixth month respectively
  recession depth was measured distance from cemento-enamel junction(CEJ) to the gingival margin, using periodontal probe at the mid-facial surface and rounded to the nearest millimeters.
root coverage | change from baseline at following surgery first, third and sixth month respectively
  Root coverage(RC) was calculated for multiple recession defects groups with a formula.
keratinized tissue thickness | change from baseline at following surgery first, third and sixth month respectively
  Keratinized tissue thickness(KTT) value was obtained from a digital caliper with the accuracy of 0.01 mm and using a 15 endodontic reamer, on mid-point localization of keratinized tissue or the alveolar mucosa, at level bottom of the gingival crevice.
keratinized tissue weight | change from baseline at following surgery first, third and sixth month respectively
  keratinized tissue weight was measured distance from the free gingival margin to the mucogingival junction, using periodontal probe at the mid-facial surface and rounded to the nearest millimeters.
clinical attachment level | change from baseline at following surgery first, third and sixth month respectively
  clinical attachment level was mesured distance from CEJ to the bottom of the gingival crevice

SECONDARY OUTCOMES:
wound healing | after surgery first, second and third week
  Wound healing was evaluated with healing index.
VAS scores for pain evaluation | after surgery first seven days
  Visual analog scale(VAS) with 100 mm was used in patient postoperative pain level for first seven days.No pain level was indicated as 0, and unbearable pain level on the VAS was also indicates as 100.

OTHER OUTCOMES:
Plaque index | change from baseline at following surgery first, third and sixth month respectively
  plaque index (Silness &Löe index) were recorded related to tooth's mean of mesial, distal, and the mid-facial surface measurements.
Gingival index | change from baseline at following surgery first, third and sixth month respectively
  Gingival index(Löe &Silness index) were recorded related to tooth's mean of mesial, distal, and the mid-facial surface measurements.
Probing pocket depth | change from baseline at following surgery first, third and sixth month respectively
  Probing pocket depth was measured distance from the gingival margin to the bottom of the gingival crevice.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Berrin Ünsal, Study Director — affiliated

IPD SHARING:
Plan to Share IPD: Undecided
there is no plan to make IPD. IPD will be formed if necessary.

REFERENCES:
- [Result] Bozkurt Dogan S, Ongoz Dede F, Balli U, Atalay EN, Durmuslar MC. Concentrated growth factor in the treatment of adjacent multiple gingival recessions: a split-mouth randomized clinical trial. J Clin Periodontol. 2015 Sep;42(9):868-875. doi: 10.1111/jcpe.12444. Epub 2015 Sep 22. PMID 26269089
- [Result] Tunaliota M, Ozdemir H, Arabaciota T, Gurbuzer B, Pikdoken L, Firatli E. Clinical evaluation of autologous platelet-rich fibrin in the treatment of multiple adjacent gingival recession defects: a 12-month study. Int J Periodontics Restorative Dent. 2015 Jan-Feb;35(1):105-14. doi: 10.11607/prd.1826. PMID 25734713
- [Result] Eren G, Atilla G. Platelet-rich fibrin in the treatment of localized gingival recessions: a split-mouth randomized clinical trial. Clin Oral Investig. 2014 Nov;18(8):1941-8. doi: 10.1007/s00784-013-1170-5. Epub 2013 Dec 22. PMID 24362634
- [Result] Jankovic S, Aleksic Z, Klokkevold P, Lekovic V, Dimitrijevic B, Kenney EB, Camargo P. Use of platelet-rich fibrin membrane following treatment of gingival recession: a randomized clinical trial. Int J Periodontics Restorative Dent. 2012 Apr;32(2):e41-50. PMID 22292152
- [Result] Jankovic S, Aleksic Z, Milinkovic I, Dimitrijevic B. The coronally advanced flap in combination with platelet-rich fibrin (PRF) and enamel matrix derivative in the treatment of gingival recession: a comparative study. Eur J Esthet Dent. 2010 Autumn;5(3):260-73. PMID 20820456
- [Result] Aroca S, Keglevich T, Barbieri B, Gera I, Etienne D. Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study. J Periodontol. 2009 Feb;80(2):244-52. doi: 10.1902/jop.2009.080253. PMID 19186964
- [Result] Del Corso M, Sammartino G, Dohan Ehrenfest DM. Re: "Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study". J Periodontol. 2009 Nov;80(11):1694-7; author reply 1697-9. doi: 10.1902/jop.2009.090253. PMID 19905939